CLINICAL TRIAL: NCT02945280
Title: Apixaban for Routine Management of Upper Extremity Deep Venous Thrombosis
Acronym: ARM-DVT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 resource allocation
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Principal Investigator, Scott C. Woller, MD, Co-Director Thrombosis Program, Intermountain Medical Center; Professor of Medicine, University of Utah School of Medicine, Intermountain Health Care, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV185-512
Record Dates: First submitted 2016-09-27; First posted 2016-10-26 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Deep Venous Thrombosis; Upper Extremity Deep Venous Thrombosis; Thrombus; Venous Thromboembolism; Deep Vein Thrombosis
Keywords: apixaban; factor Xa inhibitors; antithrombotic agent; deep vein thrombosis; upper extremity
MeSH Terms: conditions — Venous Thrombosis; Thrombosis; Venous Thromboembolism | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with acute UEDVT (Experimental): Patients will receive 10 mg PO apixaban for 7 days and then 5 mg PO for 11 weeks, for a total of 12 weeks of treatment.
  Interventions: Drug: apixaban

INTERVENTIONS:
Drug: apixaban — 12 weeks of apixaban treatment to monitor for efficacy in the prevention of VTE-related mortality
  Other Names: Eliquis

SUMMARY:
This study will assess the safety and effectiveness of a drug called apixaban for the treatment of upper extremity deep vein thrombosis (UEDVT) and clinically important bleeding. Subjects will receive apixaban 10 mg by mouth twice a day for 7 days, followed by 5 mg by mouth twice a day for a duration of 11 weeks. There will be a followup visit at 12 weeks for all participants. A total of 375 are to be enrolled.

The study drug has been approved to treat blood clots. The study drug has not been studied uniquely for the treatment of blood clots in the upper extremity however. Because it is unknown whether it is effective to treat blood clots in the upper extremity, the principal investigator cannot guarantee that there will be benefit to study subjects; however, it is hoped that the information obtained from this research study will help treat patients in the future.

DETAILED DESCRIPTION:
Background: Upper extremity deep vein thrombosis (UEDVT) constitutes approximately 10% of all DVT. A recent increase in incidence is largely secondary to the increasing use of peripherally inserted central venous catheters. Treatment for UEDVT is derived from evidence for treatment of lower extremity deep vein thrombosis (LEDVT). No evidence exists for the use of a direct oral anticoagulant (DOAC) for the treatment of UEDVT.

Population: Sequential patients identified within the Intermountain Healthcare system with UEDVT defined as the formation of thrombus within the internal jugular, subclavian, axillary, and brachial veins of the arm demonstrated by imaging.

Comparison: In the primary analysis, the principal investigator will report the rate of clinically overt objective VTE and VTE-related death in comparison to the rate reported upon literature review ("reference value in the literature"). If the confidence interval for this rate excludes the commonly accepted threshold event rate of 4%, the principal investigator will conclude that treatment with apixaban is noninferior, and therefore a clinically valid approach to treat UEDVT. As a secondary analysis, the principal investigator will compare the rate of the primary efficacy outcome and primary safety outcome with a historical control of case matched patients with UEDVT ("historical control") treated with therapy conventional (low molecular weight heparin plus warfarin) prior to the approval of DOACs.

Sample Size: A sample size of 357 patients who meet eligibility criteria was chosen so that an exact 95% confidence interval would exclude an event rate of venous thromboembolism (VTE) in the observation cohort of 4%. The principal investigator will add 5% for anticipated withdrawal to assure adequate patient enrollment in the case of patient withdrawal and enroll 375 patients.

Outcome: 90 day rate of new or recurrent objectively confirmed symptomatic venous thrombosis and VTE-related death. The primary safety outcome is major bleeding and clinically relevant nonmajor bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 years of age
* Have received no more than six (6) doses of any therapeutic anticoagulant, or intravenous and bridging heparin for longer than 72 hours
* Women must not be breastfeeding
* Receiving apixaban as administered per clinical routine (apixaban 10 mg by mouth twice daily for 7 days, followed by apixaban 5 mg twice daily for 11 weeks)
* Provide informed consent within 72 hours of receiving apixaban

Exclusion Criteria:

* Another indication for long-term anticoagulation for which no FDA approval of apixaban exists (e.g. prosthetic heart valves)
* Life expectancy of less than 6 months
* Unable to engage in reliable follow-up as per protocol
* Participating in a clinical trial or has participated in a clinical trial within the last 30 days
* Receiving concomitant dual antiplatelet therapy
* Requires aspirin dose of greater than 165 mg daily
* Intend pregnancy or breastfeeding within the next year
* Known allergy to apixaban, rivaroxaban, or edoxaban
* Active pathological bleeding.
* Any condition that at the discretion of the investigator is thought to prohibit active participation and follow-up in the trial
* UEDVT that occurs while therapeutic anticoagulation is being taken by the patient ("event on therapy")
* The patient has concomitant VTE diagnosed elsewhere except deep vein thrombosis that has its most proximal aspect in the distal veins ("isolated distal DVT")
* Any contraindication to apixaban referenced in the package insert

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Rate of recurrent symptomatic VTE and VTE-related death | 90 DAYS
  90-day rate of recurrent symptomatic venous thrombosis and venous thromboembolism-related death. If the event rate observed for venous thromboembolism (VTE) excludes 4% derived from the reference value in the literature, the principal investigator will assume noninferiority. As a secondary outcome the event rate the principal investigator observes will be compared with the historical control.
rate of major and clinically relevant nonmajor bleeding | 90 DAYS
  90-day rate of major and clinically relevant nonmajor bleeding. If the upper bound of the 95% confidence interval for event rate for the composite outcome of major bleeding and clinically relevant nonmajor bleeding excludes 13%, the principal investigator will consider apixaban as noninferior to warfarin.

SECONDARY OUTCOMES:
Patient Satisfaction | 12 weeks
  Patient satisfaction with anticoagulation will be assessed based on a standardized questionnaire called the Anti-Clot Scale (ACTS).
Patient Satisfaction | 12 weeks
  Patient satisfaction with anticoagulation will be using the Villalta scale to define and classify the severity of the post-thrombotic syndrome.
Patient Satisfaction | 12 weeks
  Patient satisfaction with anticoagulation may be assessed via a questionnaire known as the VIENES-QOL/Sym which measures the quality of life for DVT in elderly patients.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Woller, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No